CLINICAL TRIAL: NCT01599702
Title: A Prospective, Non-controlled, Safety Study of Intravenous Iron Isomaltoside 1000 (Monofer®) Administered by a High Dosing Regimen in Subjects With Inflammatory Bowel Disease (PROMISE)
Brief Title: Iron Isomaltoside 1000 (Monofer®) Administered by a High Dosing Regimen in Subjects With Inflammatory Bowel Disease
Acronym: IBD-02
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pharmacosmos A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: P-Monofer-IBD-02
Record Dates: First submitted 2012-04-25; First posted 2012-05-16 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Inflammatory Bowel Disease
Keywords: IBD; IDA; Subjects; diagnosis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Disease | interventions — iron isomaltoside 1000

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A Monofer (Experimental): Depending on the body weight, subjects in Treatment Group A will receive a total dose of 1,500 mg or 2,000 mg IV iron isomaltoside 1000 where 1,500 mg is administered as a single infusion and 2,000 mg is divided into 2 administrations: 1 administration of 1,500 mg at baseline and 1 administration of 500 mg 1 week later. All doses will be diluted in 100 ml normal saline (0.9 % sodium chloride) and administered by infusion over approximately 15 minutes.
  Interventions: Drug: Iron Isomaltoside 1000
- Group B Monofer (Experimental): Depending on the body weight, Subjects in Treatment Group B will receive a total dose of 2,500 mg or 3,000 mg IV iron isomaltoside 1000 divided into 2 administrations; 1 administration of 1,500 mg and 8 weeks later a second administration of 1,000 mg or 1,500 mg.. All doses will be diluted in 100 ml normal saline (0.9 % sodium chloride) and administered by infusion over approximately 15 minutes.
  Interventions: Drug: Iron Isomaltoside 1000

INTERVENTIONS:
Drug: Iron Isomaltoside 1000 — 1500-3000mg IV depending on HB level, sex and body weight
  Other Names: Monofer

SUMMARY:
The study is a prospective, non-controlled, open-label multi-centre pilot safety study of iron isomaltoside 1000 (Monofer®) administered to subjects with anaemia and Inflammatory Bowel Disease (IBD). Based upon haemoglobin (Hb) level, the subjects are divided into two treatment groups, A and B. Depending on the body weight, subjects in Treatment Group A will receive a total dose of 1,500 mg or 2,000 mg IV iron isomaltoside 1000 as a single infusion, whereas subjects in Treatment Group B will receive a total dose of 2,500 mg or 3,000 mg IV iron isomaltoside 1000 divided into two administrations.

DETAILED DESCRIPTION:
Subjects with a diagnosis of IBD (Crohn's disease or ulcerative colitis) and IDA ( Iron Deficiency Anaemia) with or without concomi-tant inflammation will be enrolled to receive a high dose of IV iron isomaltoside 1000.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with age ≥ 18 years
2. Subjects diagnosed with IBD either in remission or active
3. Hb < 12 g/dL for women and Hb < 13 g/dL for men
4. Subjects with a CRP above upper limit of normality must have a ferritin below 100 µg/L, whereas subjects with a CRP below or equal to upper limit of normality must have a ferritin below 30 µg/L
5. Willingness to participate after signing informed consent

Exclusion Criteria:

1. Patient judged by the physician to be in need of surgery due to Crohn´s disease or ulcerative colitis within the next 2 months
2. Anaemia predominantly caused by factors other than IDA
3. Iron overload or disturbance in utilisation of iron (e.g. haemochromatosis and haemosiderosis)
4. Known hypersensitivity to any excipients of iron isomaltoside 1000
5. History of multiple allergies
6. Decompensated liver cirrhosis and/or known chronic viral hepatitis (defined as Alanine Aminotransferase (ALAT) > 3 times upper limit of normal)
7. Acute and/or chronic infections
8. Body weight < 50 kg
9. Rheumatoid arthritis with symptoms or signs of active joint inflammation
10. Pregnancy and nursing. In order to avoid pregnancy, women have to be postmenopausal, surgically sterile, or use one of the following contraceptives during the whole study period and 5 days after the study has ended (i.e. 5 times plasma biological half-life of the investigational medicinal product): intrauterine devices and hormonal contraceptives (contraceptive pills, implants, transdermal patches, hormonal vaginal devices or injections with prolonged release)
11. Blood transfusion within the previous 12 weeks
12. Subjects with a history of asthma, allergic eczema, or other atopic allergy
13. Planned elective surgery during the study
14. Untreated Vitamin B12 or folate deficiency, defined as values below the lower reference range
15. Participation in any other clinical study within 3 months prior to Screening
16. IV iron treatment within 8 weeks prior to Screening
17. Oral iron treatment within 1 week prior to Screening
18. Erythropoiesis Stimulating Agent (ESA) treatment within 8 weeks prior to Screening
19. Any other medical condition that, in the opinion of Investigator, may cause the subject to be unsuitable for the completion of the study or place the subject at potential risk from being in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2012-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The primary objective of the study is to evaluate the safety of a high IV iron dosing regimen of iron isomaltoside 1000 in subjects with IDA secondary to IBD. | up to 16 weeks
  type and incidence of adverse drug reactions (ADRs)

SECONDARY OUTCOMES:
To evaluate the efficacy of a high IV iron dosing regimen of iron isomaltoside 1000 | up to 16 weeks
  obtain a target Hb (≥ 13 g/dL in men and ≥ 12g/dL in women)

CONTACTS AND LOCATIONS:
Locations (1):
- Pharmacosmos A/S, Hoelbaek, Denmark